CLINICAL TRIAL: NCT02092454
Title: Phase II, Multicenter, Double-Blind, Randomized, Vehicle-Controlled Study to Assess the Safety and Efficacy of Benzocaine for Pain Relief in Children Ages 2 Months to 12 Years Presenting With Acute Otitis Media
Brief Title: Study to Assess the Safety and Efficacy of Benzocaine for Pain Relief in Children Presenting With Acute Otitis Media
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otic Therapy, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OT5675
Record Dates: First submitted 2014-03-13; First posted 2014-03-20 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Pain; Acute Otitis Media
MeSH Terms: conditions — Pain; Otitis Media | interventions — Benzocaine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Benzocaine (Experimental): Topical otic solution, every 1-2 hours, for up to 3 days
  Interventions: Drug: Benzocaine
- Placebo (Placebo Comparator): Topical otic solution, every 1-2 hours, for up to 3 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Benzocaine — topical otic solution
  Arms: Benzocaine
Drug: Placebo — topical otic solution
  Arms: Placebo

SUMMARY:
To assess the clinical safety and efficacy of the Benzocaine relative to placebo in pain relief associated with acute otitis media.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ages 2 months to 12 years of age with a clinical diagnosis of AOM, and with ear pain (current episode <2 weeks duration). Baseline pain entry requires a minimum score of 4 on the FLACC or the FPS-R scale (depending on age)
* The patients must provide Institutional Review Board (IRB) approved written assent, as appropriate, which must be accompanied by an IRB approved written informed consent form (ICF) from the patient's legally acceptable representative (i.e., parent or guardian), as applicable. In addition, all patients or their legally acceptable representatives (i.e., parent or guardian) must sign a Health Insurance Portability and Accountability Act (HIPAA) authorization, if applicable
* Patients must be normally active and otherwise judged to be in good health on the basis of the medical history and a limited physical examination, as determined by the Investigator.
* Females of child bearing potential must have a negative urine human chorionic gonadotropin (hCG) pregnancy test at Visit 1

Exclusion Criteria:

* Patients with bilateral AOM, perforated tympanic membrane, history of a perforated tympanic membrane in the last 6 months, or if a perforated tympanic membrane could not be ruled out by speculum examination, impedance testing tympanometry, pneumatic otoscopy, or a Valsalva maneuver
* Patients who are subsequently diagnosed with a perforated membrane during treatment are to be discontinued immediately.
* Patients with indwelling tympanostomy tubes or draining otitis in the affected ear(s), bullous lesions, erythema of the tympanic membrane without other evidence of AOM, and patients with an anatomic defect of the ear or nasopharynx
* Complications of treated/untreated ear disease over the past 2 weeks
* Patients with comorbidity requiring antibiotic therapy, allergy to study medication, immunologic deficiency, and major medical condition(s).
* Patients with methemoglobinemia or a history of methemoglobinemia, vertigo, inherited enzyme deficiencies, impaired cardiac or respiratory functions, epilepsy, heart diseases, hypersensitivity, pyrogenic infection at or near the skin, inflamed or infected skin, dermatitis, shock, hepatic impairment, or myasthenia gravis
* Acute or chronic otitis externa
* Chronic otitis media (current episode ≥ 2 weeks)
* Patients who smoke are prohibited from participating in this study.
* Seborrheic dermatitis involving the affected external ear canal or pinna
* Any topical or systemic antibiotic received within the 14 days prior to study entry (topical antibiotics for acne will be allowed)
* Any topical drying agent or over-the-counter (OTC) therapy for otitis media received within 36 hours prior to enrollment
* Fever >102°F
* Known hypersensitivity to the study drug or similar compounds including any of the inactive ingredients
* Patients receiving medication on a chronic basis for pain (including steroidal or non-steroidal anti-inflammatory drugs)
* Use of ear drops or oral analgesics such as ibuprofen/acetaminophen within the 4 hours prior to study entry
* Use of sulfonamides, aminosalicylates, anti- cholinesterases, suxamethonium, antiarrhythmics, monoamine oxidase inhibitors, or tricyclic antidepressants
* Clinically significant mental illness (as determined by the Investigator)
* Exposure to any investigational agent within the 30 days prior to study entry
* Previous enrollment in this study
* Pregnant or lactating
* The child has a condition that the Investigator believes would interfere with the ability to provide assent (age appropriate) or comply with study instructions, or that might confound the interpretation of the study results, or put the child at undue risk

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Summed Pain Intensity Difference | 60 minutes

SECONDARY OUTCOMES:
Pain Intensity Difference | Up to 120 minutes
Comparison of pain scores from AOM-SOS and FLACC pain measurement scales in patients 2 months to 4 years old | Up to 3 days
Comparison of pain scores from VAS and FPS-R pain measurement scales in patients 5 years to 12 years old | Up to 3 days
Physician Global Evaluation | Up to 3 days
Evaluate dosing intervals with pain measurements assessed up to 120 minutes | Up to 120 minutes
Report the onset of perceptible and meaningful pain relief using patient reports and stopwatch assessments | Up to 120 minutes
  Patients will be given 2 stopwatches at the start of the study and instructed to stop one when they experience perceptible ('some') pain relief after the administration of the first dose (any change in pain intensity) and stop the other when they experience meaningful pain relief (a 'definite decrease in pain that makes them feel better')
Assess the safety and tolerability of benzocaine | Up to 3 days
  Safety will be assessed by adverse event reporting on all study days. Also, vital signs (blood pressure, pulse, temperature, and respiratory rate) and physical examinations will be assessed.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Clearwater, Florida
  - Gresham, Oregon
  - Murray, Utah